CLINICAL TRIAL: NCT05272670
Title: Taiwanese Digital Foot Self-Management Program for Older-Diabetes
Brief Title: Digital Foot Self-Management Program for Older-Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fooyin University (Other)
Responsible Party: Principal Investigator, Shu-Ming Chen, Associate Professor, Fooyin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TSMH IRB-20-084-B
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Diabetes Mellitus; Type 2 Diabetes; Glucose Metabolism Disorders; Endocrine System Diseases; Metabolic Diseases
Keywords: Digital foot self-management; Foot care self-efficacy; Self-care behaviors
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Endocrine System Diseases; Metabolic Diseases

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial will be used to examine the effectiveness of the digital foot self-management program. The outcomes included primary outcome of self-efficacy, and secondary outcomes of self-care behaviors, HbA1c and health promotion satisfaction. Participants in the intervention group will receive the digital foot self-management program in addition to routine care. The control group will receive routine care provided in diabetes clinic, including routine check-ups and foot care education.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): A 4-week digital foot self-management program will be provided to the participants in experimental group.
  Interventions: Behavioral: A digital foot self-management program
- Control group (No Intervention): The control group received routine care that are required to attend the education sessions in the diabetes clinic according to their scheduled appointments. Routine care included routine check-ups and foot care education.

INTERVENTIONS:
Behavioral: A digital foot self-management program — A 4-week digital foot self-management program based on Bandura's Self-Efficacy model. The proposed functions include checking conditions of foot, cleaning, cutting or removing corns and calluses, trimming, clipping nails, foot exercise, dietary related to foot care, foot care logs, etc. Which was developed for older adults with diabetic foot self-management by the study team. Week 1 one-hour face-to-face training session after participant recruitment and allocation. The outline session is 30 min to introduce key topics and function in the app platform, 15 min to install the app and to demonstrate the use of the app, 15min to discuss and practice. Week 2 to week 4 following phone call once per week at the end of week and LINE messages 3 times per week.by research nurse, who will encourage and monitor participant's compliance with the program at home by using the digital platform. Participants are informed that technical phone support is available during the trial.
  Arms: Experimental group

SUMMARY:
The aims of this proposed study are to evaluate the effect of a digital foot self-management program on the primary outcome of self-efficacy, and secondary outcomes of self-care behaviors, HbA1c and health promotion satisfaction for older adults with type 2 diabetes.

DETAILED DESCRIPTION:
Literature reveals the needs for diabetic foot self-management intervention programs associated with positive changes in behavior. However, lack of studies focused on measure or improve health outcomes. Promoting effective diabetic foot care strategies in community is more critical than ever during a pandemic such as COVID.

This study are to evaluate the effect of a digital foot self-management program on self-efficacy, self-care behaviors, HbA1c and health promotion satisfaction for older adults with type 2 diabetes.

The contents of the 4-week program include: using a digital platform to providing foot self-management (checking conditions of foot, cleaning, cutting or removing corns and calluses, trimming, clipping nails, foot exercise, dietary related to foot care, foot care logs, etc). A developed digital platform as a self-help foot self-management education resource. The program specifically developed for older adults with diabetes to assist and management their own feet at homes. Week 1 face-to-face training session. Week 2 to week 4 following phone call once per week and LINE messages 3 times per week.by research nurse to encourage and monitor participant's compliance with the program at home by using the digital platform.

A total of 100 older adults with type 2 diabetes will be recruited from the 5 community clinics in southern Taiwan.A computerised random number generated by an independent statistician will be used to allocate each potential participant to the control or intervention group in a one-to-one ratio. All participants will be blinded to group allocation. Participants in control group will receive routine care provided in diabetes clinic, including routine check-ups and foot care education. While participants in the intervention group received the digital foot self-management program in addition to the routine care. Data will be collected at baseline and 4 weeks from baseline for self-efficacy, self-care behaviors,health promotion satisfaction and 12 weeks from baseline for HbA1c. The digital program will be delivered by trained registered nurse. A research assistant will be blinded to study protocol, who are employed to undertake data collection.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with type 2 diabetes.
* ≧65 years.
* Possess and able to use a smart device (e.g. Samsung Galaxy, iPhone, iPad, tabletop)
* Are able to speak and comprehend Chinese

Exclusion Criteria:

* Unable to perform physical activities.
* Cognitive impairments.
* Unable to read and speak Chinese

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Foot Care Self-Efficacy Scale | 4-week
  Foot care self-efficacy was assessed using the Foot Care Self Efficacy Scale consisted of 16 items to measure individual's competence to manage foot care. Cronbach's alpha was .72. There are 16 items on the self-made scale in this study. Scored using a five-point Likert scale: "completely disagree", "slightly disagree", "no opinion", "slightly agree" and "completely agree", with a maximum score of 80 and a minimum of 16; represented higher values indicate higher foot care self-efficacy (Chen, 2005). The reliability Cronbach's alpha values were 0.82 in this study. The scale was used at baseline and week 4 for participants in both control and experimental groups.

SECONDARY OUTCOMES:
Diabetic Foot Self-Care Behavior Scale | 4-week
  Diabetic foot self-care behavior was assessed using the Diabetic Foot Self-Care Behavior Scale, a 7-item questionnaire. Cronbach's alpha was .73. The scale consists of seven questions, divided into two parts. The first part was the number of days of foot care activities and the second part was the frequency of foot care activities. On a 5-point Likert scale (never, 0 days a week= 1 point; rarely, 1-2 days a week= 2 points; sometimes, 3-4 days a week= 3 points; often, 5- 6 days a week= 4 points, 7 days a week= 5 points, with a maximum score of 35 and a minimum of 7. Represented higher scores indicate good foot self-care behavior (Chin & Huang, 2013). Internal consistency Cronbach's alpha was .89 and test-retest reliability was .92 in this study. The scale was used at baseline and 4-week for participants in both control and experimental groups.
HbA1c level | 12-week
  HbA1c level was used to present glycemic control outcome. The HbA1c level higher than 6.5% indicate worse glycemic control. The outcome was measured at baseline and at 3 months. Data were obtained from participants' medical records.
Health promotion satisfaction | 4-week
  Health promotion satisfaction will be assessed using the questionnaire of Senior Technology Acceptance Chinese version developed by Chen (Chen et al., 2020). Questionnaire consisted 4 domains: attitudinal beliefs, control beliefs, gerontechnology anxiety, health. This outcome will be measured at week 4 for participants in experimental groups.

CONTACTS AND LOCATIONS:
Overall Officials: Fooyin University, Principal Investigator — Nursing Department
Locations (1):
- Fooyin University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen SM, Lin HS, Atherton JJ, MacIsaac RJ, Wu CJ. Effect of a mindfulness programme for long-term care residents with type 2 diabetes: A cluster randomised controlled trial measuring outcomes of glycaemic control, relocation stress and depression. Int J Older People Nurs. 2020 Sep;15(3):e12312. doi: 10.1111/opn.12312. Epub 2020 Feb 26. PMID 32103635
- [Background] Wu CJ, Atherton JJ, MacIsaac RJ, Courtney M, Chang AM, Thompson DR, Kostner K, MacIsaac AI, d'Emden M, Graves N, McPhail SM. Effectiveness of the cardiac-diabetes transcare program: protocol for a randomised controlled trial. BMC Health Serv Res. 2017 Feb 2;17(1):109. doi: 10.1186/s12913-017-2043-4. PMID 28153000